CLINICAL TRIAL: NCT04955015
Title: Associations of Carotid Plaque Characteristics With Brain Perfusion and Cognitive Function in Patients Undergoing CEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019292
Record Dates: First submitted 2021-06-29; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Atherosclerosis of Artery; Carotid Endarterectomy
Keywords: atherosclerosis; carotid endarterectomy; perfusion; cognition
MeSH Terms: conditions — Atherosclerosis | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients: patients with caotid atherosclerosis refering to carotid endarterectomy
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid endarterectomy — patients with carotid atherosclerosis refering to CEA

SUMMARY:
Stroke is one of the leading causes of death and disability-adjusted life-years worldwide. Carotid high-risk atherosclerotic plaques are considered to be one of the major sources of ischemic stroke. The present study aimed to investigate the relationship of carotid plaque characteristics with brain perfusion and cognitive function in patients undergoing carotid endarterectomy.

DETAILED DESCRIPTION:
Cerebrovascular disease is the first cause of death and adult disability in China. More than 75% of the patients in China have ischemic cerebrovascular disease, and about 33.3% of them have ipsilateral extracranial carotid stenosis. One of the main causes of carotid stenosis is atherosclerosis. Atherosclerotic plaques can be divided into two types: stable plaques and vulnerable plaques. Vulnerable plaque has the tendency to rupture, prone to thrombosis and rapid progression of dangerous plaque. Its pathological characteristics are mainly as follows: thin fibrous cap (or fibrous cap has been broken), large lipid nucleus, massive hemorrhage in plaque, rich in inflammatory cells, abundant neovascularization and plaque surface calcification. Vulnerable plaque is the main cause of stroke. At present, high-resolution magnetic resonance imaging combined with multi sequence is one of the best methods to evaluate carotid artery stenosis, which is helpful to analyze plaque characteristics.

At present, the main treatment methods of carotid artery stenosis are: carotid endarterectomy (CEA) and carotid angioplasty with stenting (CAS). Large scale multicenter prospective randomized trials and meta-analysis have established CEA as the gold standard for the treatment of carotid arerosclerotic stenosis.

Studies have shown that the ipsilateral cerebral perfusion is continuously decreased due to carotid artery stenosis, and CEA operation can relieve the vascular stenosis and improve the cerebral perfusion. However, the relationship between cerebral perfusion improvement after CEA and the quantitative characteristics of vulnerable plaque is still lack of sufficient evidence. Vascular cognitive impairment is closely related to the progress of carotid stenosis. The main mechanisms are microemboli formation, white matter injury and central nervous function decline caused by long-term chronic hypoperfusion. The formation and continuous hypoperfusion of microemboli further increase the burden of white matter disease. Studies have shown that the visual spatial executive ability, naming ability, attention ability and abstract profile ability of patients after CEA are significantly improved. However, there is still insufficient evidence about the relationship between the MRI features of vulnerable carotid plaques and the improvement of cognitive function after CEA.

We hope to achieve the following goals: 1) to explore the associations between carotid vulnerable plaque characteristics and cerebral perfusion in patients undergoing CEA; 2) to explore the associations between the characteristics of vulnerable carotid plaques and cognitive function in patients undergoing CEA.

ELIGIBILITY:
Inclusion Criteria:

1. Over 30 years old;
2. The patients with symptomatic (>50%) or asymptomatic carotid stenosis (> 70%) measured by computed tomography angiography (CTA) or B-mode ultrasonography
3. CEA operation will be performed in our hospital.

Exclusion Criteria:

1. The history of CEA operation in the last 3 months;
2. Diseases (AF, valve diseases, etc.) that may cause cardiac thrombosis;
3. Contraindications of MR examination (vascular stent implantation, pacemaker, metal or magnetic plants in vivo, claustrophobia, etc.) were found;
4. Contraindications of contrast agents: such as renal failure, iodine or gadolinium contrast agent allergy;
5. Having heart or respiratory failure;
6. Serious consciousness disorder (coma, etc.);
7. Brain tumor;
8. Acute cerebral hemorrhage;
9. Pregnant women or planned pregnancies in the past 2 years;
10. Who does not agree to sign the informed consent.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with carotid atherosclerosis refering to CEA in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
brain perfusion | From preoperative to 24 months after operation (CEA)
  perioperative brain perfusion and changes of brain perfusion in patients underging CEA
cognitive function | From preoperative to 24 months after operation (CEA)
  perioperative cognitive function and cognitive changes in patients underging CEA

CONTACTS AND LOCATIONS:
Overall Officials: Huishu Yuan, Dr., Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China